CLINICAL TRIAL: NCT01356147
Title: Pilot Study of Dornase Alfa (Pulmozyme) Therapy for Acquired Ventilator Associated Infection in Preterm and Late Preterm Infants in the Neonatal Intensive Care Unit
Brief Title: Dornase Alfa Therapy for Ventilator Associated Lung Infections in the Neonatal Intensive Care Unit (NICU)
Acronym: PVAIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Melissa Scala, Assistant Professor of Pediatrics, Department of Neonatology, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Z4962s
Record Dates: First submitted 2011-03-29; First posted 2011-05-19 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-07

CONDITIONS: Pulmonary Infections
Keywords: ventilator associated pulmonary infections
MeSH Terms: interventions — dornase alfa

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham placebo (Sham Comparator): No therapy will be given to placebo arm. Respiratory therapist will shield infant from view and nebulize saline solution into incubator rather than into ventilator circuit.
  Interventions: Drug: Placebo
- Dornase alfa (Active Comparator): Dornase alfa 2.5 mg nebulized endotracheally every 12 hours for 7 days or until extubation
  Interventions: Drug: Dornase alfa

INTERVENTIONS:
Drug: Dornase alfa — 2.5 mg nebulized endotracheally every 12 hours for 7 days or until extubation
  Other Names: Pulmozyme
  Arms: Dornase alfa
Drug: Placebo — No therapy will be given to placebo arm
  Other Names: Sham therapy
  Arms: Sham placebo

SUMMARY:
To evaluate the effect of Dornase alfa on preterm and late preterm neonates with ventilator associated pulmonary infections. Dornase alfa has been effective in the treatment of pulmonary infections in patients with cystic fibrosis by aiding mucus clearance. The bacteria causing pulmonary infections in cystic fibrosis patients is similar to those infecting preterm infants. The investigators expect that dornase alfa therapy will improve recovery from ventilator associated pulmonary infections in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* infants less than 38 weeks gestation and over 7 days of age
* infants with a ventilator associated pulmonary infection, defined as intubated infants who have moderate to heavy White Blood Cells (WBCs) on tracheal aspirate, organisms on tracheal aspirate gram stain, a positive endotracheal tube culture, a chest x-ray with infiltrate, consolidation or atelectasis, an increase in oxygen (FiO2) requirement and whom the clinical team decides to treat with systemic antibiotic therapy

Exclusion Criteria:

* Extremely ill infants not expected to survive
* Critically ill infants requiring high frequency ventilation
* Infants with congenital pneumonia
* Infants with congenital malformations of the respiratory system (e.g. Congenital diaphragmatic hernia, cystic adenomatoid malformation or tracheo-esophageal fistula) Cyanotic congenital heart disease, chromosomal abnormalities and infants with a positive newborn screen for cystic fibrosis

Ages: 7 Days to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2011-05; Primary Completion 2015-01 (Actual); Study Completion 2017-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Georgetown University Hospital NICU, Washington D.C., District of Columbia
  - Georgetown University Hospital, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medstar Georgetown University Hospita NICU patients recruited from May 2012 to november 2014
Pre-assignment Details: No enrolled participants were excluded prior to assignment to groups
Period: Overall Study
Arm/Group | Sham Placebo | Dornase Alfa
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Placebo | Dornase Alfa | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 6 | 11
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: days] | 29 [18 to 39] | 33 [18 to 68] | 31 [18 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percent Reduction in Oxygen Requirement From Baseline
Description: Change in required supplemental oxygen from baseline or time to extubation from mechanical ventilation
Time Frame: First week of treatment or extubation
Measure: Mean (Full Range); unit: percentage FiO2
Arm/Group | Sham Placebo | Dornase Alfa
Number analyzed (Participants) | 5 | 6
percentage FiO2 | 5.4 [-2 to 23] | 16.5 [-4 to 73]

2. Secondary Outcome: Elimination of White Blood Cells and Bacteria From Tracheal Aspirate
Description: Number of infants with Tracheal aspirate WBC present on review of smear at end of therapy Bacterial load judged on presence of positive or negative culture in Tracheal aspirate
Time Frame: During first week of treatment or until extubation whichever is earlier
Measure: Number; unit: participants
Arm/Group | Sham Placebo | Dornase Alfa
Number analyzed (Participants) | 5 | 6
participants | 1 | 4

3. Secondary Outcome: Number of Infants Requiring Ventilator Support
Description: number of infants extubated during treatment/sham
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Sham Placebo | Dornase Alfa
Number analyzed (Participants) | 5 | 6
participants | 1 | 0

ADVERSE EVENTS:
Time Frame: During 7 day period of drug or sham treatment then throughout NICU admission
Arm/Group | Sham Placebo | Dornase Alfa
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No